CLINICAL TRIAL: NCT02132182
Title: A Canine/ Human Translational Model of Phenotypic and Functional Differences Between Monocytes in Patients With and Without Sarcoma
Brief Title: Monocyte Phenotypic and Functional Differences
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050745
Record Dates: First submitted 2014-04-21; First posted 2014-05-07 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples (~15 to 20 mls) will be obtained from 90 humans over 3 years presenting to Duke with osteosarcoma. Only patients who would normally have blood drawn as part of standard care will be included. Research blood will be in addition to what is normally collected. Samples will be de-identified and then transferred to researchers as NC State's College of Veterinary Medicine. These researchers will use the samples to perform a CBC and evaluate monocyte phenotype and function. These results will be compared to published historical normal values for healthy human monocytes. This data will also be compared with canine data already gathered.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients newly diagnosed with osteosarcoma: Blood draw
  Interventions: Biological: Blood draw

INTERVENTIONS:
Biological: Blood draw — The patient population for this study will be comprised of individuals who present to clinic with newly diagnosed osteosarcoma with or without infection and without known metastasis to the lung. These patients would have a standard-of-care blood draw. For the study we will be drawing an additional 15-20mL of blood (no additional needle stick).

SUMMARY:
The purpose of this study is to identify phenotypic (cell surface receptor expression) and functional differences in monocyte populations in humans with osteosarcoma as compared to published historical data on normal human monocyte values.

The biologic similarity between canine and human osteosarcoma makes it a disease model that holds promise for translational research possibilities. The phenotypic and functional differences the investigators expect to find in canine and human monocytes between normal and osteosarcoma subjects in this pilot work will allow us to launch a program of investigations to further their understanding as to what characteristics are associated with improved survival in canine and human osteosarcoma. Such data will represent the foundation upon which the investigators can plan future investigations designed to exploit the potential anti-tumor capabilities of monocytes and macrophages in canine and human osteosarcoma.

DETAILED DESCRIPTION:
Research on canine osteosarcoma lends itself well to comparative studies of osteosarcoma in humans because dogs develop spontaneous tumors which are similar to human cancers with the added benefit of frequently being more prevalent1. Osteosarcoma is diagnosed in more than 8000 dogs every year, and it affects mostly middle-aged to older dogs.2 The majority (75%) of canine osteosarcoma occurs in the appendicular skeleton.3 Osteosarcoma is diagnosed in 1-3 million humans every year, and is a disease primarily of those between 10 and 25 years old. Human osteosarcoma also occurs primarily in the appendicular skeleton, and like dogs, is most often found in the metaphyses of long bones. Pulmonary metastasis is the most common site of spread in dogs and humans, and is usually the cause of death in patients that have undergone standard of care therapy (surgical resection of tumor, chemotherapy).4 The reported median survival times for canine osteosarcoma have plateaued with no notable improvements in the last 20 years, despite attempts at various permutations of adjunctive chemotherapy.5,6,7 Targeting metastatic disease will be the key to improving survival in both canine and human osteosarcoma.

Interestingly, there is one arena in which median survival times in osteosarcoma have been extended - patients who develop infections after limb-spare surgery have been observed to double their median survival time. Lascelles et al. noted that infected dogs were half as likely to die, half as likely to develop metastasis, and these survival effects were due to a delay in metastasis rather than control of local tumor recurrence.8 A similar phenomenon of increased survival in infected human osteosarcoma patients has been observed. Jeys et al.reported that the 10-year survival rate in humans was significantly better in infected limb-spares: 84.5% in the infected patients versus 62.2% in the non-infected patients.9 An upregulation of antitumor immunity has been postulated to be potentially responsible for the favorable survivals in the face of an infection in dogs and humans. Characterization of the phenotype and function of circulating canine and human monocytes in normal subjects, and in osteosarcoma subjects with and without an infection will be crucial in furthering their understanding of how these cells are involved in the pathogenesis and potential suppression of osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for evaluation of osteosarcoma of the appendicular skeleton
* Patient is 6years or older at time of visit
* Patients do not need to be eligible for surgery
* Patients may have known infection related to osteosarcoma and its treatment (ex. surgical wound infection)
* Patients who would normally have a blood draw as part of their standard care

Exclusion Criteria:

* Patients younger than 10 years of age
* Patients who are unwilling/unable to undergo blood draw
* Patients with known infection unrelated to osteosarcoma or its treatment
* Patients with known systemic immune-mediated disease including but not limited to lymphoma, AIDS/HIV, Lupus, etc.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population for this study will be comprised of individuals who present to clinic with newly diagnosed osteosarcoma with or without infection and without known metastasis to the lung. Potential subjects will be 10 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Variations in the intensity of cell surface receptor expression | 1 day
  We will characterize the phenotypic differences demonstrated by variations in cell surface receptor expression, such as CCR2, CCR7 and CD32, between normal monocytes and monocytes in osteosarcoma patients.

CONTACTS AND LOCATIONS:
Overall Officials: William Eward, MD, DVM, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States